CLINICAL TRIAL: NCT05376124
Title: Clinical Characteristics, Natural Outcome and Treatment Optimization of Refractory Hepatitis B: a Open Label, Prospective, Multi-center Cohort Study
Brief Title: Clinical Characteristics, Natural Outcome and Treatment Optimization of Refractory
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2021CRF-006
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-10

CONDITIONS: Hepatitis B, Chronic; Virus Diseases
Keywords: HBV; Refractory hepatitis B; Clinical characteristics; Natural outcome; nucleoside analog
MeSH Terms: conditions — Hepatitis B, Chronic; Virus Diseases; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- original therapy: ETV 0.5mg/ day or TDF 300mg/ day or TAF 25mg/ day continued the original regimen (ETV 1.0mg/ day or TDF 300mg/ day or TAF 25mg/ day), Oral treatment lasted 48 weeks ②TDF 300mg/ day plus ETV 0.5mg/ day on initial treatment continued with the original regimen (TDF 300mg/ day plus ETV 0.5mg/ day) and oral therapy for 48 weeks ③TAF 25mg/ day plus ETV 0.5mg/ day as initial treatment continued the original regimen (TAF 25mg/ day plus ETV 0.5mg/ day) for 48 weeks of oral therapy
  Interventions: Other: original therapy
- rescue therapy: TDF 300mg/ day +ETV 1.0mg/ day or TAF 25mg/ day +ETV 1.0mg/ day, oral treatment for 48 weeks.
  Interventions: Other: rescue therapy

INTERVENTIONS:
Other: original therapy — * Patients on ETV 0.5mg/ day or TDF 300mg/ day or TAF 25mg/ day continued the original regimen (ETV 1.0mg/ day or TDF 300mg/ day or TAF 25mg/ day), Oral treatment lasted 48 weeks ②Patients who received TDF 300mg/ day plus ETV 0.5mg/ day on initial treatment continued with the original regimen (TDF 300mg/ day plus ETV 0.5mg/ day) and oral therapy for 48 weeks ③Patients who received TAF 25mg/ day plus ETV 0.5mg/ day as initial treatment continued the original regimen (TAF 25mg/ day plus ETV 0.5mg/ day) for 48 weeks of oral therapy
  Groups: original therapy
Other: rescue therapy — TDF 300mg/ day +ETV 1.0mg/ day or TAF 25mg/ day +ETV 1.0mg/ day, oral treatment for 48 weeks.
  Groups: rescue therapy

SUMMARY:
Refractory hepatitis B is to point to although standard application nucleoside (acid) analogue treatment undertakes primary treatment and two strengthen treatment, but existence is persistent viremia. Currently, there is no consensus on salvage therapy for patients who remain virus-positive after a second round of antiviral therapy. This is the first multicenter, prospective, parallel controlled, open-label cohort study to compare the efficacy and safety of TDF/TAF combined with ETV1.0mg regimen versus continuation of the original regimen in the treatment of refractory hepatitis B.

DETAILED DESCRIPTION:
Refractory sex hepatitis B is to point to although standard application nucleoside (acid) analogue treatment undertakes first treat and 2 strengthen treat cure, but existence is persistent viraemia. These patients have active liver inflammation and are at high risk for progression to cirrhosis or primary liver cancer due to persistent virus-positive symptoms. Therefore, it is of great significance to find an effective antiviral program for refractory hepatitis B to reduce the fatality rate of hepatitis B in China. At present, the guidelines recommend that patients with drug resistance to Entecavir (ETV) be treated with tenofovir fumarate (TDF) or propofol tenofovir fumarate (TAF), and clinical studies in China have confirmed that increased dosage of entecavir to 1.0mg can be used as the treatment of drug resistance to entecavir. TDF and TAF resistant patients can be treated with entecavir 0.5mg. However, currently there is no consensus on salvage treatment for patients who remain virus-positive after a second round of antiviral therapy. Previous studies have shown that TDF/TAF combined with ETV 1.0mg as a rescue regimen has no obvious adverse drug reactions. This is the first multicenter, prospective, parallel controlled, open-label cohort study to compare the efficacy and safety of TDF/TAF combined with ETV 1.0mg regimen versus continuation of the original regimen in the treatment of refractory hepatitis B. Meanwhile, long-term outcomes of refractory hepatitis B patients, such as survival, cirrhosis and primary liver cancer, were observed. In addition, the effects of refractory hepatitis B virus strain, host and other clinical characteristics on the antiviral efficacy of nucleoside (acid) analogue were compared with those of patients with initial treatment and secondary enhancement of nucleoside (acid) analogue response. The results of this study are expected to provide a new perspective for the treatment of refractory hepatitis B and provide direct evidence for the formulation of guidelines for the diagnosis and treatment of chronic hepatitis B in China and even internationally.

ELIGIBILITY:
Inclusion Criteria:

* (1) The diagnostic criteria of chronic hepatitis B: HBsAg and/or HBV DNA positive for more than 6 months; (2) Conforming to the definition of refractory hepatitis B (3) Aged between 18 and 70 (including 18 and 70); (4) Willing to accept treatment and sign informed consent.

Exclusion Criteria:

* (1) Pregnant women or lactating women; (2) with active HEPATITIS A, hepatitis C, and hepatitis D (in hospitals where conditions permit), hepatitis E and/or HIV infection; (3) Decompensated cirrhosis (Child-Pugh score 6); (4) Symptoms and signs of hepatocellular carcinoma, AFP> Patients with 100ng/ml of AFP would be excluded, but patients whose AFP remained stable (increased by less than 10%) for more than 3 months prior to the trial could be enrolled in patients whose liver tumors were excluded by liver imaging if AFP> 20ng/mL but 100ng/mL can be selected; (5) In addition to viral hepatitis, other history or evidence related to chronic liver disease (such as hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposure, thalassemia); (6) a history of serious mental illness, especially depression severe mental illness is defined as at least 3 months before the above treatment dose antidepressant or antipsychotic drug treatment of severe depression or psychosis, or there are any medical history: once for attempted suicide was hospitalized due to mental illness, or had a disability due to mental illness; (7) a history of severe seizures or current use of anticonvulsants; (8) a history of chronic lung disease related to functional limitations; (9) A history of severe heart disease (NYHA grade III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmia requiring continued treatment, unstable angina or other important cardiovascular disease); (10) patients who are participating in other trials or have been treated with the study drug in the 12 weeks prior to screening; (11) Patients with a history of allergy to ETV, TDF and TAF; In addition to the above exclusion criteria, patients who meet any of the contraindications in the experimental drug description; (12) Unable or unwilling to provide informed consent or comply with the requirements of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory hepatitis B in January 2022 to January 2023 of The First Affiliated Hospital of Xi 'an Jiaotong University、The Second Affiliated Hospital of Xi 'an Jiaotong University、 Xijing Hospital Air Force Medical University 、Tang-du Hospital 、Shaanxi Provincial People's Hospital Xi 'an Central Hospital、 Ankang Central Hospital 、Yan 'an University Affiliated Hospital、 Hanzhong 3201 Hospital Weinan Central Hospital 、The First Affiliated Hospital of Shandong Medical University、Wuhan Union Hospital、The First Affiliated Hospital of Zhengzhou University.
  All patients were required to sign written informed consent before enrollment
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative HBV-DNA conversion | 48weeks
  Negative HBV-DNA conversion at 48 weeks of treatment
Liver hardness measurement | 3 years
  3-year liver hardness measurement (LSM value)
Hepatocellular carcinoma | 3 years
  Incidence and survival of hepatocellular carcinoma.

SECONDARY OUTCOMES:
virology indicators | 48weeks
  virology indicators: quantitative hbv-dna;
Biochemical indexes | 3 years
  Biochemical indexes: ALT level;
Immunological indicators | 3 years
  Immunological indicators: HBsAg level and HBsAg disappearance HBeAg serological conversion;
Drug-related adverse reactions | 3 years
  Drug-related adverse reactions

OTHER OUTCOMES:
Strain mutation indicators | 1year,2years and 3years
  Strain mutation indicators: High-throughput sequencing was used to detect the presence of 5 preS1 deletion mutations at 1, 2, and 3 years after baseline treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yingren Zhao, Principal Investigator — Department of Infectious Diseases, The First Affiliated Hospital of Xi'an Jiaotong University
Locations (13):
- China (13):
  - Ankang Central Hospital, Ankang
  - Hanzhong 3201 Hospital, Hanzhong
  - Qianfhan Hospital, Jinan
  - Weinan Central Hospital, Weinan
  - Wuhan Union Hospital, Wuhan
  - Department of Infectious Diseases, The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Shaanxi Provincial People's Hospital, Xi'an
  - Tang-Du Hospital, Xi'an
  - Xi'an Central Hospital, Xi'an
  - Xijing hospital of air force Medical University, Xi'an
  - Yan'an University Affiliated Hospital, Yan’an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou